CLINICAL TRIAL: NCT07286227
Title: Assessment of Left Ventricular Function Before Decannulation in Cardiopulmonary Bypass Surgeries: Comparison of the Cardiac Surgeon's Visual Estimation and Transesophageal Echocardiography
Brief Title: Assement of Left Ventricular Function Before Decannulation in Cardiac Surgery :Visual Estimation vs TEE
Acronym: LVFuncTee
Status: Not yet recruiting | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed E Aydin, DOÇENT.DR, Ataturk University
Other Study IDs: B.30.2.ata.0.01.00/767
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cardiopulmonary Bypass Surgery; Left Ventricular Dysfunction
Keywords: Transesophageal Echocardiography; Left Ventricular Ejection Fraction; Visual Estimation; Eyeballing Method; Cardiac Surgery; Ejection Fraction Assessment; Intraoperative Monitoring; Decannulation; Cardiopulmonary Bypass
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiopulmonary Bypass Cohort: Patients undergoing elective cardiac surgery with cardiopulmonary bypass (CABG, valve surgery, or aortic procedures). During the decannulation phase, left ventricular function will be assessed visually by the cardiac surgeon (eyeballing method) and objectively by intraoperative transesophageal echocardiography (TEE). No additional intervention is performed. Both evaluations are part of standard intraoperative monitoring. Data will be recorded simultaneously to compare the accuracy and agreement between visual estimation and TEE-derived ejection fraction.
  Interventions: Diagnostic Test: Intraoperative Left Ventricular Function Assessment

INTERVENTIONS:
Diagnostic Test: Intraoperative Left Ventricular Function Assessment — Left ventricular function will be assessed during the decannulation phase of cardiopulmonary bypass using two diagnostic methods: (1) visual estimation of ventricular contractility by the cardiac surgeon (eyeballing) and (2) objective measurement using intraoperative transesophageal echocardiography (TEE). No experimental procedure, medication, or additional intervention will be applied. Both assessments are part of standard intraoperative monitoring in cardiac surgery. Data from both methods will be collected simultaneously to compare accuracy, agreement, and diagnostic performance.
  Other Names: Visual Estimation (Eyeballing); Transesophageal Echocardiography (TEE)

SUMMARY:
This study aims to evaluate the diagnostic performance of the cardiovascular surgeon's visual estimation of LV function before decannulation following cardiopulmonary bypass, using TEE results as the reference standard.

DETAILED DESCRIPTION:
The fundamental rationale for conducting this study is that the moment of decannulation after cardiopulmonary bypass (CPB) represents one of the most critical stages in cardiac surgery in terms of patient outcomes. At this stage, inadequate left ventricular (LV) function (dysfunction) can lead to severe hemodynamic deterioration, increased complications, and a higher risk of mortality. Therefore, accurately and rapidly assessing LV function just before separation from CPB is of vital importance. Although Transesophageal Echocardiography (TEE) is currently the most reliable and objective method, it requires specialized equipment, training, and time. On the other hand, experienced cardiac surgeons often make a visual estimation based on the observable physical appearance of the heart (such as its color, contractility, and fullness), relying on their many years of experience. This visual assessment is extremely fast and practical; however, it is subjective, and its reliability has not been clearly established scientifically.

Thus, the primary rationale for this study is to fill this gap in the scientific literature and determine how well the surgeon's quick, experience-based visual estimation aligns with the objective findings of TEE, the gold-standard method.

The main objective of the study is to evaluate the diagnostic performance of the cardiovascular surgeon's visual estimation of LV function before decannulation following cardiopulmonary bypass, using TEE results as the reference standard. In other words, it aims to statistically determine the agreement between the surgeon's practical visual assessment and the objective measurements provided by TEE, thereby offering a scientific basis for clinical decision-making by revealing the sensitivity and specificity limits of the surgeon's estimation, particularly in detecting critical conditions such as severe dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Scheduled for elective cardiac surgery requiring cardiopulmonary bypass (CABG, valve surgery, or aortic surgery)
* ASA physical status III-IV
* Able and willing to provide written informed consent
* Suitable for intraoperative transesophageal echocardiography (TEE)

Exclusion Criteria:

* Emergency surgery
* Known severe preoperative left ventricular dysfunction (EF < 30%)
* Significant arrhythmias (e.g., atrial fibrillation)
* Preoperative requirement for mechanical circulatory support (e.g., IABP)
* Contraindications to TEE (esophageal pathology, bleeding risk, strictures)
* Inability to provide informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery requiring cardiopulmonary bypass at a single tertiary university hospital. The study population consists of individuals receiving CABG, valve surgery, or aortic surgery who meet eligibility criteria and undergo routine intraoperative TEE monitoring. Participants represent a typical clinical population of moderate-to-high surgical risk (ASA III-IV).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Agreement Between Surgeon Visual Estimation and TEE-Derived Left Ventricular Ejection Fraction | During the decannulation phase of cardiopulmonary bypass (intraoperative period)
  This outcome evaluates the level of agreement between the cardiac surgeon's visual estimation (eyeballing) of left ventricular systolic function and the ejection fraction measured by intraoperative transesophageal echocardiography (TEE). Agreement will be quantified using statistical measures such as Cohen's kappa coefficient and correlation coefficients. Visual estimation categories (e.g., normal, moderately reduced, severely reduced) will be compared with corresponding TEE-derived EF classifications.

SECONDARY OUTCOMES:
Diagnostic Accuracy of Surgeon Visual Estimation for Detecting Reduced Left Ventricular Function | During the decannulation phase of cardiopulmonary bypass (intraoperative period)
  This outcome measures the diagnostic performance of the surgeon's visual estimation in identifying reduced left ventricular systolic function, using TEE-derived ejection fraction as the reference standard. Sensitivity, specificity, positive predictive value, negative predictive value, and overall accuracy will be calculated for detecting clinically significant systolic dysfunction (e.g., EF < 30% or EF < 40%).
Prediction of Postoperative Hemodynamic Support Requirement | From intraoperative decannulation through 24 hours postoperatively
  This outcome evaluates whether the surgeon's intraoperative visual assessment of left ventricular function predicts the need for postoperative hemodynamic support. Outcomes include the requirement for intra-aortic balloon pump (IABP), return to cardiopulmonary bypass, or initiation of high-dose inotropic therapy during or after separation from bypass.
Correlation Between Quantitative TEE Measurements and Surgeon Visual Estimation | During the decannulation phase of cardiopulmonary bypass
  This outcome examines the correlation between TEE-derived quantitative parameters (ejection fraction, end-diastolic volume, end-systolic volume) and the categorical visual estimation provided by the cardiac surgeon (normal, moderately reduced, severely reduced). Correlation coefficients (Pearson or Spearman) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Enes Aydın, Principal Investigator, Principal Investigator — Ataturk University Department of Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding IPD sharing has not yet been finalized. If data sharing is pursued in the future, it will involve de-identified datasets and will comply with institutional and ethical regulations.

REFERENCES:
- [Background] Kim H. Weaning from cardiopulmonary bypass. Korean J Anesthesiol. 2013 Jun;64(6):487-8. doi: 10.4097/kjae.2013.64.6.487. No abstract available. PMID 23814646
- [Background] Abazid RM, Abohamr SI, Smettei OA, Qasem MS, Suresh AR, Al Harbi MF, Aljaber AN, Al Motairy AA, Albiela DE, Almutairi BM, Sakr H. Visual versus fully automated assessment of left ventricular ejection fraction. Avicenna J Med. 2018 Apr-Jun;8(2):41-45. doi: 10.4103/ajm.AJM_209_17. PMID 29682476
- [Background] Metkus TS, Thibault D, Grant MC, Badhwar V, Jacobs JP, Lawton J, O'Brien SM, Thourani V, Wegermann ZK, Zwischenberger B, Higgins R. Transesophageal Echocardiography in Patients Undergoing Coronary Artery Bypass Graft Surgery. J Am Coll Cardiol. 2021 Jul 13;78(2):112-122. doi: 10.1016/j.jacc.2021.04.064. Epub 2021 May 3. PMID 33957241
- [Result] Bayram E, Gulcu O, Aksu U, Aksakal E, Birdal O, Kalkan K. Evaluating the Association Between the Three Different Ejection Fraction Measurement Techniques and Left Ventricle Global Strain. Eurasian J Med. 2018 Oct;50(3):173-177. doi: 10.5152/eurasianjmed.2018.17409. PMID 30515038